CLINICAL TRIAL: NCT06889467
Title: Validation of Liquid Biopsy Assay of EBUS-TBNA Supernatant Fluid for Diagnosing Lung Cancer: A Feasibility Study
Brief Title: Liquid Biopsy Assay of EBUS-TBNA Supernatant Fluid for Diagnosing Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Ori Wand, Head, Division of Pulmonary Medicine, Barzilai Medical Center
Other Study IDs: BRZ-0076-22
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Non Small Cell Lung Cancer; Non Small Cell Lung Cancer (NSCLC); Lung Cancer (NSCLC); Lung Cancer - Non Small Cell; Pulmonary Nodule
Keywords: Endobronchial ultrasound; Endobronchial ultrasound transcbronchial needle aspiration; EBUS; EBUS-TBNA; staging; lung cancer; non small cell lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — supernatant fluid from EBUS-TBNA procedures peripheral blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adults with high suspicion for NSCLC: Pdult (age ≥18 years) patients with high suspicion for NSCLC with thoracic lymph nodes involvement (per clinical judgement and imaging studies), planned for an EBUS-TBNA procedure, will be recruited. Only subjects with a negative EBUS-TBNA results (no evidence of lymph node involvement by tumor according to histology) who will require surgical resection of the thoracic lymph nodes will comprise the final study group

SUMMARY:
Background and aim: Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) is the gold standard of lung cancer staging, yet up to 15% of procedures produce inadequate samples for definite diagnosis or staging. In such cases, more invasive surgical procedures are usually considered. Fluid collected during EBUS-TBNA is centrifuged to produce a pellet for cell block histopathological examination , while the supernatant is usually discarded. It has been demonstrated that this supernatant can provide material for next generation sequencing (NGS) mutation analysis using liquid biopsy (LB) technics when the procedure yielded positive results (tumor cells were demonstrated in the aspirate).

We wish to assess whether LB NGS of the supernatant may provide data regarding lymph nodes involvement in non-small cell lung cancer (NSCLC) in cases with a negative EBUS-TBNA evaluation (no tumor cell identified in the aspirate).

Methods: A prospective feasibility study which will recruit participants with high suspicion for thoracic lymph nodes involvement in NSCLC who will be subjected to EBUS-TBNA. The final study group will comprise of 10 subjects with a negative EBUS-TBNA evaluation (no tumor cell detected) who will require surgical resection of the thoracic lymph nodes.

EBUS-TBNA collected fluid will be centrifuged and separated. Cellular pellets will undergo cytological and histopathological evaluation, including tissue NGS, as usual. Cell-free DNA will be extracted from the supernatant and will undergo separate LB NGS targeted to genes frequently mutated in NSCLC. We will assess the concordance between the positivity of supernatant NGS and surgical lymph nodes staging, and the concordance between supernatant NGS and blood NGS.

Expected results: We expect high concordance between surgical lymph nodes staging and supernatant NGS, that is, genetic mutations would be identified by the supernatant NGS in subjects with lymph nodes involvement by tumor, and not in those without it.

Importance to Medicine: NSCLC is the leading cause of cancer mortality. Improving the effectiveness of EBUS-TBNA may reduce the need for additional invasive procedures, increase accuracy and reduce turnaround time of specimens.

DETAILED DESCRIPTION:
Background Lung cancer is the leading cause of cancer deaths. In particular, non-small cell lung cancers (NSCLC) accounts for over 80% of cases. Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) is the first-choice procedure for staging of NSCLC, as it allows a low-risk, minimally invasive histopathological tumor diagnosis, and provides adequate material for immunohistochemistry staining and molecular testing. During the procedure, thoracic lymph nodes are sampled under endobronchial sonographic guidance. However, 10-15% of EBUS-TBNA does not yield adequate cytological material for precise diagnosis, staging, or further testing. This may result from sampling errors, low quality or quantity of collected material, or abundance of necrosis. In those cases, further invasive surgical procedures such as mediastinoscopy or thoracoscopy may be considered to complete the staging determination.

Next generation sequencing (NGS) of tumor cells is recommended to identify molecular alterations to select targeted therapies and improve outcomes. When tissue samples are limited or non-diagnostic, NGS can also be performed on peripheral blood or other body fluids, such as malignant pleural effusions and EBUS-TBNA supernatant, by liquid biopsy (LB) technics. Molecular profiling of peripheral blood by LB is highly concordant with NGS of tissue biopsies, the same mutations are detected by both methods, and is thus gaining an increasing popularity in the management of patients with NSCLC. LB can provide a molecular characterization when tissue quality or quantity is not sufficient, identify possible therapeutic targets when such are not detected by tissue NGS, and guide further treatment in cases of disease progression. LB NGS of EBUS-TBNA supernatant was assessed in several small-scale studies, which found good concordance with NGS of tissue biopsies and peripheral blood, improved failure rates, and possibly reduced costs and turnaround times. Those studies included supernatant from positive procedures only, that is, procedures in which tumor cells were identified from EBUS-TBNA samples. Currently, LB NGS cannot ascertain (or rule-out) lymph nodes involvement in tumor development, and thus cannot contribute to the staging process.

This study aim is to preliminary assess whether LB NGS from the supernatant could contribute to identifying lymph nodes involvement in subjects diagnosed with NSCLC, but determined as negative for lymph nodes involvement by EBUS-TBNA.

The study hypothesis is that there is an excellent correlation between LB NGS from EBUS-TBNA supernatant and tumor involvement of the lymph nodes, even when such involvement is unrecognized by EBUS-TBNA cytology.

Study Objectives General Aim To preliminary assess whether LB NGS of the supernatant may be indicative of lymph node involvement in patients with non-small cell lung cancer (NSCLC) in whom no tumor cells have been identified in the aspirate (false negative).

Specific Aims

1. To assess the concordance between the positivity of supernatant LB NGS and surgical lymph nodes staging in subjects with a negative EBUS-TBNA evaluation (no tumor cell detected) who will require surgical resection of the thoracic lymph nodes.
2. To assess the concordance between LB NGS of the supernatant and NGS of surgical tumor specimens.
3. To assess the concordance between LB NGS of the supernatant and LB NGS from peripheral blood.

Methods This is a prospective feasibility study. The primary outcome will be the concordance between the results of EBUS-TBNA supernatants NGS (positive vs. negative for any mutation commonly associated with NSCLC) and the final pathological staging following surgery (positive vs. negative thoracic lymph nodes involvement). Secondary exploratory outcome will be the concordance between genetic alterations detected by comprehensive tissue NGS and those detected by supernatant LB, cell-free DNA NGS, and the concordance between peripheral blood and supernatant LB NGS.

Inclusion Criteria:

1. Ten adult (age ≥18 years) patients with high suspicion for NSCLC with thoracic lymph nodes involvement (per clinical judgement and imaging studies), planned for an EBUS-TBNA procedure, will be recruited.
2. Subjects with negative EBUS-TBNA results (no evidence of lymph node involvement by tumor according to histology) who will require surgical resection of the thoracic lymph nodes will comprise the final study group.

Exclusion Criteria:

1. Subjects unable or not willing to provide informed consent for study participation.
2. Subjects in whom NSCLC will ultimately be ruled out.
3. Subjects who will not require surgical resection of thoracic lymph nodes, or who will not undergo such procedure in our Medical Center for any reason.

Sample Size:

10 participants will be recruited for this feasibility study. This should allow detection of a significant agreement (Cohen's Kappa) of >0.55, with 80% power and type I error (alpha) of 0.05.

Measured Variables:

Collected data will include:

* Age
* Gender
* Smoking history
* Past medical history, co-morbidities, and medications
* Imaging results and radiological staging
* EBUS-TBNA report, including lymph nodes size and structure, number, and location of sampled nodes
* Surgery reports
* Final surgical pathology and staging
* NGS of tumor tissue from surgical specimens
* LB NGS from EBUS-TBNA supernatant
* Treatment decisions

Study Procedures:

Participants will undergo EBUS-TBNA procedures under moderate sedation, as commonly practiced. During the procedures, suspicious thoracic lymph nodes will be sampled using sonographic guidance. EBUS-TBNA needle and syringe rinse fluid will be collected in tubes containing 30ml of CytoLyt (Hologic, Marlborough, Massachusetts). Samples will be centrifuged at 1200 RPM for 10 minutes, the supernatant will be poured into another tube, and the cell pellet will be fixed in formalin and embedded in paraffin as a cell block, for standard cytopathological workup. The supernatant (which is usually discarded) will be stored at 4°C until surgical resection of the lymph nodes will be recommended by a Tumor Board.

DNA and RNA will be extracted from formalin-fixed and paraffin-embedded (FFPE) tissue for NGS using Oncomine™ Comprehensive Assay Plus for therapeutic decisions as generally practiced. For the subjects in the final study group, cell-free DNA will be extracted from the supernatant samples and NGS will be performed using Oncomine™ Pan-Cancer Cell-Free Assay, and also from peripheral blood, according to manufacturer recommendations and as previously described. Both assays can detect a wide spectrum of genetic mutations which are typically associated with NSCLC. All extractions, sequencing, analysis, and calculation will be performed in the Pathology Laboratory of Barzilai University Medical Center.

Statistical Analysis:

Descriptive statistics will include mean and medians with standard deviations and range, absolute numbers, and percentages. Agreement between tests will be calculated using Cohen's Kappa statistic.

ELIGIBILITY:
Inclusion Criteria:

* adult (age ≥18 years) patients with high suspicion for NSCLC with thoracic lymph nodes involvement (per clinical judgement and imaging studies), planned for an EBUS-TBNA procedure
* Subjects with negative EBUS-TBNA results (no evidence of lymph node involvement by tumor according to histology) who will require surgical resection of the thoracic lymph nodes will comprise the final study group

Exclusion Criteria:

1. Subjects unable or not willing to provide informed consent for study participation.
2. Subjects in whom NSCLC will ultimately be ruled out.
3. Subjects who will not require surgical resection of thoracic lymph nodes, or who will not undergo such procedure in our Medical Center for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo surgical resection of thoracic lymph nodes for NSCLC following an EBUS-TBNA procedure which was negative for tumor cell in the thoracic lymph nodes.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
EBUS-TBNA NGS accuracy | 1 year
  The concordance between the positivity of supernatant LB NGS and surgical lymph nodes staging in subjects with a negative EBUS-TBNA evaluation (no tumor cell detected) who will require surgical resection of the thoracic lymph nodes

SECONDARY OUTCOMES:
Accuracy of EBUS-TBNA and tissue NGS | 1 year
  The concordance between EBUS-TBNA liquid biopsy NGS of the supernatant and NGS of surgical tumor specimens
peripheral blood and EBUS-TBNA concordance | 1 year
  The concordance between liquid biopsy NGS of the EBUS-TBNA supernatant and liquid biopsy NGS from peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilai University Medical Center, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: Yes
Will be provided following reasonable request from the PI
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 31 Dec 2025 for 2 years
Access Criteria: additional data will be provided following reasonable request from the PI